CLINICAL TRIAL: NCT02753309
Title: A Randomized Study of Rapamycin Combined With Intravesical BCG in Patients With Non-muscle Invasive Bladder Cancer
Brief Title: A Study of Rapamycin Combined With Intravesical BCG in Patients With Non-muscle Invasive Bladder Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC20160162H
Record Dates: First submitted 2016-04-18; First posted 2016-04-27 (Estimated); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Bladder Cancer
Keywords: BCG; Rapamycin
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Rapamycin 0.5mg (Active Comparator): Subject will take Rapamycin (Sirolimus) 0.5mg once daily for approximately 28 days
  Interventions: Drug: Sirolimus
- Rapamycin 2.0mg (Active Comparator): Subject will take Rapamycin (Sirolimus) 2.0mg once daily for approximately 28 days
  Interventions: Drug: Sirolimus
- Control (No Intervention): Subject will be apart of the control group and won't take the study drug being tested

INTERVENTIONS:
Drug: Sirolimus
  Other Names: Rapamycin; Rapamune
  Arms: Rapamycin 0.5mg; Rapamycin 2.0mg

SUMMARY:
This study is looking at the effects of Sirolimus (Rapamycin) on BCG-specific immunity during treatment of non-muscle invasive bladder cancer (NMIBC) with maintenance BCG.

DETAILED DESCRIPTION:
This study will evaluate change from baseline in gamma-delta T cell numbers and function and Ag85 peptide-specific T cell responses following treatment.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically) proven diagnosis of non-muscle invasive (Ta, Tis or T1) bladder cancer
* In their treating physician's opinion is a good candidate for BCG therapy
* Be able to give informed consent
* Be age 18 or older
* Not be in an immunosuppressed state (e.g. HIV, use of chronic steroids)
* Not have active, uncontrolled infections
* Not be on agents known to alter rapamycin metabolism significantly
* Not have a reported history of liver disease (e.g. cirrhosis)
* Not have a prior history of non-bladder cancer unless the cancer is clinically stable and not requiring active treatment except basal cell carcinoma or squamous cell carcinoma of the skin.
* Not pregnant, or taking effective contraception before rapamycin therapy, during therapy and for 12 weeks after discontinuation of therapy.

Exclusion Criteria:

* Have muscle-invasive (≥T2) bladder cancer
* Unable to give informed consent
* Age < 18
* Immunosuppressed state (e.g. HIV, use of chronic steroids)
* Active, uncontrolled infections
* On agents known to alter rapamycin metabolism significantly
* Another cancer requiring active treatment (except basal cell carcinoma or squamous cell carcinoma of the skin)
* Patients at risk of pregnancy who are unwilling or unable to take effective contraception before rapamycin therapy, during therapy, and for 12 weeks after discontinuation of therapy.
* Individuals with a reported history of liver disease (e.g. cirrhosis)
* Individuals who are not a good candidate for BCG in their treating physician's opinion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-06; Primary Completion 2019-12-01 (Actual); Study Completion 2021-03-02 (Actual)

PRIMARY OUTCOMES:
Percentage change in systemic (whole blood) gamma-delta T cells frequency | 4 weeks and 3 months after therapy
  Change will be evaluated by comparing percentage increase or decrease following rapamycin or control (no therapy) against baseline measures
Percentage change in systemic (whole blood) gamma-delta T cell proliferation in response to BCG-specific antigens | 4 weeks and 3 months after therapy
  Change will be evaluated by comparing percentage increase or decrease following rapamycin or control (no therapy) against baseline measures
Percentage change in systemic (whole blood) Ag85 peptide-specific CD4 and CD8 T lymphocytes measured using human IFN-gamma release. | 4 weeks and 3 months after therapy
  Change will be evaluated by comparing percentage increase or decrease following rapamycin or control (no therapy) against baseline measures

CONTACTS AND LOCATIONS:
Overall Officials: Robert Svatek, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

REFERENCES:
- [Derived] Ji N, Mukherjee N, Reyes RM, Gelfond J, Javors M, Meeks JJ, McConkey DJ, Shu ZJ, Ramamurthy C, Dennett R, Curiel TJ, Svatek RS. Rapamycin enhances BCG-specific gammadelta T cells during intravesical BCG therapy for non-muscle invasive bladder cancer: a randomized, double-blind study. J Immunother Cancer. 2021 Mar;9(3):e001941. doi: 10.1136/jitc-2020-001941. PMID 33653802